CLINICAL TRIAL: NCT02232971
Title: Treatment of Hypoglycemia With Glucagon Among Patients With Type 1 Diabetes Mellitus
Brief Title: Treatment of Low Blood Sugar With Glucagon Among Patients With Type 1 Diabetes
Acronym: GluST1
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Hvidovre University Hospital (Other)
Collaborators: The Novo Nordic Foundation (Other); University of Copenhagen (Other)
Responsible Party: Principal Investigator, Ajenthen Ranjan, MD, PhD student, Hvidovre University Hospital
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: GluST1_2014; 2014-002267-15 (EudraCT Number); H-1-2014-041 (Other: The National Committee on Health Research Ethics)
Record Dates: First submitted 2014-08-29; First posted 2014-09-05 (Estimated); Last update posted 2015-03-25 (Estimated); Status verified 2015-03

CONDITIONS: Diabetes Mellitus, Type 1
Keywords: glucagon; insulin pump; artificial pancreas; closed-loop
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — Glucagon; Glucagon-Like Peptide 1

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Placebo (Placebo Comparator): Isotonic Saline
  Interventions: Other: Isotonic saline solution
- Glucagon 0.1 mg (Experimental): GlucaGen(r) 0.1 mg administration
  Interventions: Drug: Glucagon
- Glucagon 0.2 mg (Experimental): GlucaGen(r) 0.2 mg administration
  Interventions: Drug: Glucagon
- Glucagon 0.3 mg (Experimental): GlucaGen(r) 0.3 mg administration
  Interventions: Drug: Glucagon

INTERVENTIONS:
Drug: Glucagon — Glucagon is given in three different doses according to three research days.
  Other Names: GlucaGen (r); Disp. no. 2514; Novo Nordisk A/S; Novo Allé; 2880 Bagsværd
  Arms: Glucagon 0.1 mg; Glucagon 0.2 mg; Glucagon 0.3 mg
Other: Isotonic saline solution — Placebo
  Other Names: Natriumklorid isotonisk "SAD"; D.sp.no. 6733; Amgros I/S; Dampfærgevej 22; Postbox 2593; 2100 København Ø
  Arms: Placebo

SUMMARY:
Background: Patients with type 1 diabetes (T1D) need a lifelong supply of external insulin and are advised to aim for near-normalization of blood glucose levels through intensive insulin therapy. We propose a new approach for achieving treatment goals in T1D: the combined use of insulin and glucagon, i.e. dual-hormone treatment.Only recently the prospect of treating patients with soluble glucagon has arisen and thus studies of low dose glucagon treatment of mild hypoglycemia are needed to determine whether there is clinical rationale for dual-hormone treatment of T1D.

Aim: The purpose of this clinical study is to investigate the glycemic response to subcutaneous glucagon administration during mild hypoglycemia in T1D patients treated with insulin pump. Different glucagon doses are applied to determine the most appropriate dose for future dual-hormone treatment of T1D.

Methods: A clinical, randomized, single blinded, crossover study will be conducted. Eight T1D patients treated with insulin pump are studied on four days. All patients are in good metabolic control (HbA1c < 7.5%), C-peptide negative and with hypoglycemia awareness. On each study day, hypoglycemia is induced with subcutaneously insulin and afterward treated with a single subcutaneous dose of glucagon. The study procedures are identical on all days except from the administered dose of glucagon (day 1: placebo, day 2: 100 ug, day 3: 200 ug, day 4: 300 ug). All patients are blinded for the glucagon dose and carry out the four days in random order.

Endpoints: The present study focuses primarily on the dose related plasma glucose response of glucagon; secondary on the duration of the hyperglycemic effect of glucagon and tertiary the glucagon effect on catecholamine, cortisol, growth hormone, free fatty acids and triglycerides.

The study will be conducted from august 2014.

ELIGIBILITY:
Inclusion Criteria:

* Males and females aged 18-65 years
* Diagnosed with type 1 diabetes > 3 years
* HbA1c < 58 mmol/mol
* No appearance of autonome neuropathy
* Body mass index (BMI) between 20-25 kg/m2
* Remained hypoglycemic awareness
* Insulin pump treatment > 1 year

Exclusion Criteria:

* Allergic to glucagon or lactose
* Pregnancy, breast-feeding, intention of becoming pregnant, or not using adequate contraception
* Any disease or condition which would interfere with the subject's safety
* Use of a medication that significantly impacts glucose metabolism

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Estimated)
Dates: Start 2014-09; Primary Completion 2015-01 (Actual); Study Completion 2015-07 (Estimated)

PRIMARY OUTCOMES:
Maximum plasma glucose response | Plasma glucose measured every five minutes after administration

SECONDARY OUTCOMES:
Duration of hyperglycemic effect of glucagon | Plasma glucose is measured every five minutes. Time period is two -three hours after glucagon administration

OTHER OUTCOMES:
Plasma Catecholamine | Measured at 0, 5, 10, 15, 30, 45, 60, 90, 120,180, 240 minutes after glucagon administration
Plasma free fatty acids | Measured at 0, 5, 10, 15, 30, 45, 60, 90, 120,180, 240 minutes after glucagon administration
Plasma Beta-Hydroxybutyric acid | Measured at 0, 5, 10, 15, 30, 45, 60, 90, 120,180, 240 minutes after glucagon administration
Plasma Glucagon | Measured at 0, 5, 10, 15, 30, 45, 60, 90, 120,180, 240 minutes after glucagon administration
Serum Growth hormone | Measured at 0, 5, 10, 15, 30, 45, 60, 90, 120,180, 240 minutes after glucagon administration
Serum Cortisol | Measured at 0, 5, 10, 15, 30, 45, 60, 90, 120,180, 240 minutes after glucagon administration
Serum Insulin (Novorapid) | Measured at 0, 5, 10, 15, 30, 45, 60, 90, 120,180, 240 minutes after glucagon administration
Adverse reaction: Stomach pain | One time before and after insulin administration. One time before glucagon administration. After glucagon administration at T=15 min., T=60 min., T=120 min., T=240 min.
  Visual analog scale
Adverse reaction: Headache | One time before and after insulin administration. One time before glucagon administration. After glucagon administration at T=15 min., T=60 min., T=120 min., T=240 min.
  Visual Analog scale
Adverse Reaction: Vertigo | One time before and after insulin administration. One time before glucagon administration. After glucagon administration at T=15 min., T=60 min., T=120 min., T=240 min.
  Visual analog scale
Adverse reaction: Nausea | One time before and after insulin administration. One time before glucagon administration. After glucagon administration at T=15 min., T=60 min., T=120 min., T=240 min.
  Visual analog scale
Adverse reaction: Hunger | One time before and after insulin administration. One time before glucagon administration. After glucagon administration at T=15 min., T=60 min., T=120 min., T=240 min.
  Visual analog scale
Plasma triglycerides | Measured at 0, 5, 10, 15, 30, 45, 60, 90, 120,180, 240 minutes after glucagon administration

CONTACTS AND LOCATIONS:
Overall Officials: Ajenthen Ranjan, MD, Principal Investigator — Hvidovre University Hospital; Signe Schmidt, MD, PhD, Study Director — Hvidovre University Hospital; Kirsten Nørgaard, MD, DMSc, Study Chair — Hvidovre University Hospital; Sten Madsbad, Prof, DMSc, Study Chair — Hvidovre University Hospital; Jens J Holst, Prof, DMSc, Study Chair — University of Copenhagen
Locations (1):
- Hvidovre University Hospital, Hvidovre, Denmark